CLINICAL TRIAL: NCT00411580
Title: A 52-week, Multi-center, Randomized, Double-blind, Placebo-controlled, Time-lagged, Parallel Group Study in Patients With Mild to Moderate Alzheimer's Disease (AD) to Investigate the Safety, Tolerability and Aß-specific Antibody Response Following Three Subcutaneous Injections of CAD106
Brief Title: Safety and Tolerability Study in Patients With Mild to Moderate Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCAD106A2101
Record Dates: First submitted 2006-12-13; First posted 2006-12-14 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Alzheimer's Disease
Keywords: Mild, moderate Alzheimer's Disease (AD), Aß-specific antibody, CAD106
MeSH Terms: conditions — Alzheimer Disease; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): CAD106
  Interventions: Biological: CAD106
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CAD106
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study will evaluate the safety and tolerability and Aß-specific antibody response of CAD106 in patients with mild to moderate Alzheimer's Disease.

Patients also had a 2 year follow-up to assess disease progression where no drug was administered.

ELIGIBILITY:
Inclusion Criteria:

* males and/or females patients between 50 to 80 years of age (both inclusive).
* female patients must be without childbearing potential (post-menopausal or surgically sterilized).
* diagnosis of dementia of the Alzheimer's type according to the DSM-IV criteria (Diagnostic and Statistical Manual of Mental Disorders, 4th edition).
* mild to moderate AD as confirmed by Mini-Mental State Exam score of 16 to 26 (both inclusive) at screening.
* able to provide written informed consent and having a responsible caregiver that can provide written assent prior to study participation. For patients who have been declared mentally incompetent, a legal representative will need to provide informed consent on their behalf.

Exclusion Criteria:

* previously participated in an AD vaccine study and received active treatment
* history or presence of an active autoimmune and/or cerebrovascular disease
* history or presence of seizures, with an acute or chronic inflammation
* clinically relevant atopic condition, who suffer from an other neurodegenerative disease and/or psychiatric disorders (with the exception of successfully treated depression)
* immunosuppressive treatment including systemic steroids
* obtained a vaccination (e.g. against influenza) within 4 weeks before the first study drug injection
* advanced, severe, progressive or unstable disease that might interfere with the safety of the patient
* started treatment with psychotropic medication within 3 months (4 weeks for SSRIs and other newer antidepressants without anticholinergic properties) prior to randomization with the exception of mild hypnotic drugs (e.g. zolpidem, zopiclone, oxazepam) and low doses of neuroleptic drugs (e.g. up to 2 mg risperidone).

Patients, who are on stable treatment with cholinesterase-inhibitors (ChEIs) and/or memantine for at least 3 months, and/or with SSRIs and/or other newer antidepressants (without anticholinergic properties) for at least 4 weeks before randomization, can be included into the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Tolerability/safety assessments (physical/neurol.exam., ECG, vital signs, standard and special immunological laboratory evaluations, MRIs, EEGs, AE/SAE monitoring). | at multiple timepoints including but not limited to screening, baseline, and through the end of the study to Week 52.
Antibody titers (IgM and IgM titers against amyloid and carrier protein). | at multiple timepoints including but not limited to baseline and through the end of the study to Week 52

SECONDARY OUTCOMES:
Immune response, cognitive and functional assessments | at multiple timepoints including but not limited to baseline and through the end of the study to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Principal Investigator — Investigator site
Locations (2):
- Sweden (2):
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Stockholm

REFERENCES:
- [Derived] Winblad B, Andreasen N, Minthon L, Floesser A, Imbert G, Dumortier T, Maguire RP, Blennow K, Lundmark J, Staufenbiel M, Orgogozo JM, Graf A. Safety, tolerability, and antibody response of active Abeta immunotherapy with CAD106 in patients with Alzheimer's disease: randomised, double-blind, placebo-controlled, first-in-human study. Lancet Neurol. 2012 Jul;11(7):597-604. doi: 10.1016/S1474-4422(12)70140-0. Epub 2012 Jun 6. PMID 22677258